CLINICAL TRIAL: NCT00951444
Title: A Randomized Phase II Study of Gemcitabine and Carboplatin With or Without MK-0646 as First-Line Therapy in Advanced Squamous Non-Small Cell Lung Carcinoma
Brief Title: Gemcitabine Hydrochloride and Carboplatin With or Without MK-0646 as First-Line Therapy in Treating Patients With Stage IIIB or Stage IV Non-Small Cell Lung Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was not activated.
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: N0823; NCCTG-N0823; CDR0000650608 (Registry Identifier: PDQ (Physician Data Query)); NCI-2011-01957 (Registry Identifier: CTRP (Clinical Trials Reporting System))
Record Dates: First submitted 2009-08-01; First posted 2009-08-04 (Estimated); Last update posted 2016-07-06 (Estimated); Status verified 2016-07

CONDITIONS: Lung Cancer
Keywords: adenosquamous cell lung cancer; squamous cell lung cancer; recurrent non-small cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — dalotuzumab; Carboplatin; Gemcitabine

ARMS (2):
- Arm I (Experimental): Patients receive gemcitabine hydrochloride IV over 30 minutes on days 1 and 8, carboplatin IV over 30 minutes on day 1, and MK-0646 IV over 60 minutes on days 1, 8, and 15. Treatment repeats every 21 days for 4 courses in the absence of disease progression or unacceptable toxicity. After 4 courses, patients with stable disease or partial or complete response may then receive MK-0646 alone on days 1 and 15. Treatment with MK-0646 repeats every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: dalotuzumab; Drug: carboplatin; Drug: gemcitabine hydrochloride
- Arm II (Active Comparator): Patients receive gemcitabine hydrochloride and carboplatin as in arm I. Treatment repeats every 21 days for 4 courses in the absence of disease progression or unacceptable toxicity. Patients may crossover to arm upon disease progression.
  Interventions: Drug: carboplatin; Drug: gemcitabine hydrochloride

INTERVENTIONS:
Biological: dalotuzumab — Given IV
  Arms: Arm I
Drug: carboplatin — Given IV
Drug: gemcitabine hydrochloride — Given IV

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as gemcitabine hydrochloride and carboplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as MK-0646, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. It is not yet known whether gemcitabine hydrochloride and carboplatin are more effective when given together with or without MK-0646 in treating patients with non-small cell lung cancer.

PURPOSE: This randomized phase II trial is studying how well gemcitabine hydrochloride and carboplatin work when given together with or without MK-0646 as first-line therapy in treating patients with stage IIIB or stage IV non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To assess and compare the progression-free survival of patients with stage IIIB or IV squamous cell non-small cell lung cancer treated with gemcitabine hydrochloride and carboplatin with vs without MK-0646 as first-line therapy.

Secondary

* To assess and compare the objective tumor response rate in patients treated with these regimens.
* To assess and compare the duration of response in patients with objective tumor response treated with these regimens.
* To assess and compare the time to progression and time to treatment failure in patients treated with these regimens.
* To assess and compare the 1-year overall survival of patients treated with these regimens.
* To assess and compare the clinical toxicities of these regimens in these patients.
* To compare the quality of life of patients treated with these regimens.

Tertiary

* To collect blood and tumor specimens for future evaluation of pharmacogenetic and proteomic markers of tumor response and toxicity to therapy.
* To assess the relationship between ht-SNPs in genes that mediate chemosensitivity/resistance to gemcitabine hydrochloride (e.g. ribonucleotide reductase) and IGF1R pathway genes.
* To bank paraffin-embedded tissue blocks/slides for future histochemistry evaluation and DNA extraction as part of ongoing research for NCCTG lung studies.

OUTLINE: This is a multicenter study. Patients are stratified according to prior adjuvant therapy, neoadjuvant therapy, or chemoradiotherapy (yes vs no), and ECOG performance status (0 vs 1 vs 2). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive gemcitabine hydrochloride IV over 30 minutes on days 1 and 8, carboplatin IV over 30 minutes on day 1, and MK-0646 IV over 60 minutes on days 1, 8, and 15. Treatment repeats every 21 days for 4 courses in the absence of disease progression or unacceptable toxicity. After 4 courses, patients with stable disease or partial or complete response may then receive MK-0646 alone on days 1 and 15. Treatment with MK-0646 repeats every 28 days in the absence of disease progression or unacceptable toxicity.
* Arm II: Patients receive gemcitabine hydrochloride and carboplatin as in arm I. Treatment repeats every 21 days for 4 courses in the absence of disease progression or unacceptable toxicity. Patients may crossover to arm I upon disease progression.

Blood and tissue samples may be collected for pharmacogenetics and further laboratory analysis.

Quality of life is assessed at baseline and periodically during study.

After completion of study treatment, patients are followed up periodically for up to 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed squamous cell non-small cell lung cancer (NSCLC)

  * Squamous histology mixed with other NSCLC component (e.g. adenosquamous) allowed

    * No mixed histology with small cell component
* Stage IV disease
* Candidate for palliative chemotherapy
* Measurable disease, defined as ≥ 1 lesion whose longest diameter can be accurately measured as ≥ 2.0 cm by chest X-ray OR as ≥ 1.0 cm by CT scan, CT component of a PET/CT scan, or MRI

  * If the sole site of disease was previously irradiated, there must be evidence of disease progression at that site
* No symptomatic, untreated, or uncontrolled CNS metastases
* Concurrent enrollment on NCCTG-N0392 required

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Life expectancy ≥ 12 weeks
* ANC ≥ 1,500/μL
* Platelet count ≥ 100,000/μL
* Hemoglobin ≥ 9 g/dL
* Total bilirubin normal (< 3.0 mg/dL for patients with Gilbert syndrome)
* ALT and AST ≤ 2.5 times upper limit of normal (ULN)
* Alkaline phosphatase ≤ 5 times ULN
* Creatinine clearance ≤ 1.2 times ULN OR calculated creatinine clearance ≥ 60 mL/min
* Fasting glucose < 120 mg/dL
* HbA1c ≤ 7%
* INR < 1.5 OR PT/PTT normal (patients receiving anticoagulation therapy with an agent such as warfarin or prophylactic-dose heparin are eligible provided the patient meets the above criteria at the patient's stable dose of anticoagulants)
* QTc < 450 msec and no conduction abnormalities (e.g., heart block) on EKG

  * Isolated premature ventricular or atrial conduction beats allowed
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Willing and able to comply with study
* Willing to return to NCCTG participating center for follow-up
* Willing to provide blood samples as required by study
* Able to complete questionnaire(s) alone or with assistance
* No clinically significant infection
* No significant traumatic injury within the past 4 weeks
* No symptomatic, untreated, or uncontrolled seizure disorder
* No uncontrolled diabetes mellitus, defined as fasting blood glucose ≥ 120 mg/dL on 2 consecutive measurements (taken ≤ 2 weeks apart) or by patient's clinical history
* No other uncontrolled illness including, but not limited to, any of the following:

  * Ongoing or active infection
  * Significant pulmonary symptoms at baseline due to disease
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia
  * Psychiatric illness/social situation that would limit compliance with study requirements
* No second primary malignancy, except for any of the following:

  * Carcinoma in situ of the cervix
  * Nonmelanomatous skin cancer
  * Other malignancy that was diagnosed and definitively treated ≥ 5 years ago with no subsequent evidence of recurrence
  * History of low-grade (Gleason score ≤ 6) localized prostate cancer, even if diagnosed within the past 5 years
  * Stage I breast cancer that was treated within the past 5 years
* No HIV-positivity and no history of chronic hepatitis B or C (regardless of viral load)
* No evidence or history of bleeding diathesis or coagulopathy

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior chemotherapy for advanced lung cancer, except neoadjuvant therapy, adjuvant therapy, or chemoradiotherapy for lung cancer administered > 12 months ago
* More than 12 months since prior gemcitabine hydrochloride, cisplatin, or carboplatin
* More than 12 months since prior immunotherapy or biologic therapy
* At least 1 week since prior gamma knife radiosurgery for brain metastases or palliative radiotherapy for skeletal metastases and recovered
* At least 2 weeks since prior whole-brain radiotherapy for CNS metastases and recovered
* More than 2 weeks since other prior radiotherapy
* No prior radiotherapy to ≥ 25% of bone marrow
* More than 2 weeks since prior minor surgery*
* More than 4 weeks since prior major surgery (e.g., laparotomy)*
* No other concurrent anticancer drugs or therapy
* No concurrent therapeutic anticoagulation

  * Prophylactic anticoagulation (i.e., low-dose warfarin) of venous or arterial access devices allowed provided the requirements for PT, INR, or PTT are met
* Concurrent radiotherapy for symptom palliation allowed
* Concurrent megestrol acetate for appetite allowed NOTE: *Insertion of a vascular access device is not considered major or minor surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | Up to 5 years

SECONDARY OUTCOMES:
Overall survival | Up to 5 years
Response rate, defined as complete or partial response noted as the objective status on 2 consecutive evaluations at least 6 weeks apart | Up to 5 years
Time to disease progression | Up to 5 years
Time to treatment failure | Up to 5 years
Duration of response | Up to 5 years
Toxicity according to NCI CTCAE v.3 | Up to 5 years
Quality of life using single-item Linear Analogue Self Assessment (single-item LASA) and single-item measure for fatigue at baseline, at the end of courses 2 and 4, and at the end of treatment | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Grace K. Dy, MD, Study Chair — Roswell Park Cancer Institute